CLINICAL TRIAL: NCT03443882
Title: Bioavailability of Astaxanthin Formulations
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Algatechnologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 01 2018 ver1
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Astaxanthin formulation #1 (Active Comparator): capsules
  Interventions: Dietary Supplement: Astaxanthin
- Astaxanthin formulation #2 (Active Comparator): tablets
  Interventions: Dietary Supplement: Astaxanthin
- Astaxanthin formulation #3 (Active Comparator): powder
  Interventions: Dietary Supplement: Astaxanthin
- Astaxanthin formulations (Experimental): fast condition
  Interventions: Dietary Supplement: Astaxanthin

INTERVENTIONS:
Dietary Supplement: Astaxanthin — an oral dose form

SUMMARY:
Bioavailability of dietary supplement formulations in healthy volunteers after a single oral dose.

DETAILED DESCRIPTION:
Comparison of the bioavailability of 3 formulations with astaxanthin in healthy volunteers after single dose

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed an informed consent form and who meet all of the following entrance criteria may be enrolled in this clinical trial: Generally, healthy men and women who are 21 to 50 years of age, inclusive, at the baseline visit.

Exclusion Criteria:

* 1. Are unwilling to follow the procedures of the trial, such as making visits or having their blood drawn.

  2. Have unintentionally lost or gained 10 or more kg of body weight in the last 3 months; 3. Have an acute illness (such as a severe cold or flu) or have been hospitalized within the past month for certain conditions; 4. Have severe co-morbid disease including cardiac, pulmonary, renal, hepatic, carotid, peripheral vascular disease, stroke, neurological, clotting disorders or active cancer; 5. Taking chronic drugs which interfere with lipids metabolism (statins or similar) 6. Consume alcohol at an elevated level (Defined as consumption of more than 10 standard alcoholic drinks per week. A standard alcoholic drink is defined as one bottle/can of beer or one glass of wine equals one portion of hard liquor).

  7. Consume carotenoids as food supplements. 8. Have a Body Mass Index (BMI) of less than 17 or greater than 35 m/kg2; 9. Have participated in a clinical trial in the past 4 weeks; 10. Have any disease or condition that in the investigator's opinion compromises the integrity of the clinical trial or the safety of the subject; 11. Smokers 12. Pregnant woman

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
plasma level | 0-48 hr
  astaxanthin in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Bitzur, MD, Principal Investigator — Bert W. Strassburger Lipid Center, Sheba Medical Center, Tel Hashomer
Locations (1):
- Bert W. Strassburger Lipid Center, Sheba Medical Center,, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No